CLINICAL TRIAL: NCT03563495
Title: Clinical, Volumetric and Densitometric Evaluation of Tissue Engineered (TE) Constructs for Secondary Alveolar Cleft Reconstruction (Short Term Randomized Controlled Clinical Trial)
Brief Title: Tissue Engineered Constructs for Alveolar Cleft Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Kadry, principal investigator at Oral & Maxillofacial Surgery department, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: MSCs in alveolar cleft repair
Record Dates: First submitted 2018-05-26; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Cleft Lip and Palate
Keywords: tissue engineering.; stem cells.; autogenous grafts.
MeSH Terms: conditions — Cleft Lip | interventions — osteovit

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tissue engineered group (Active Comparator): autogenous bone marrow derived and cultured stem cells loaded on collagen matrix was implanted in the alveolar cleft in the study group (1st arm)
  Interventions: Other: tissue engineered group
- autogenous bone graft group (Active Comparator): autogenous cortico-cancellous bone graft harvested from the anterior iliac crest was implanted in the alveolar cleft of the control group (2nd arm)
  Interventions: Procedure: autogenous bone graft group

INTERVENTIONS:
Other: tissue engineered group — cultured and bone marrow derived autologous mesenchymal stem cells, loaded on collagen matrix (Osteovit)
  Other Names: BM-MSCs on collagen matrix (Osteovit)
  Arms: tissue engineered group
Procedure: autogenous bone graft group
  Arms: autogenous bone graft group

SUMMARY:
Description of the research question

In children undergoing unilateral alveolar cleft reconstruction, would stem cells carried on collagen scaffold provide bone of a good quality and quantity if compared to autogenous bone grafting?

Objective of the study:

• Research hypothesis

The tissue engineered constructs will provide sufficient bone of a good quality and quantity if compared to autogenous bone graft in children undergoing unilateral alveolar cleft reconstruction.

* The objectives

The primary objective:

Assessment of bone volume (quantity) which will be provided by tissue engineered constructs compared to that provided by autogenous bone for maxillary alveolar cleft reconstruction.

The secondary objective:

Assessment of bone density (quality) which will be provided by tissue engineered constructs compared to that provided by autogenous bone for maxillary alveolar cleft reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Children with maxillary unilateral alveolar clefts requiring reconstruction
* Children free from any systemic disease that may affect normal healing of bone
* Children in an age range (8-14) year.

Exclusion criteria

* Bilateral alveolar clefts.
* Cleft lip or palate not including the alveolus.
* Immunocompromized patients.
* Children who undergone previous bone grafting procedure for the alveolar cleft

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in the bone volume at the grafted alveolar cleft site from the immediate postoperative to 6 months | Immediate postoperative and after 6 months
  Measuring the bone volume on CT scan

SECONDARY OUTCOMES:
Assessment of changes in the bone density at the grafted alveolar cleft site from the immediate postoperative to 6 months | Immediate postoperative and after 6 months
  Measuring the bone density on CT scan